CLINICAL TRIAL: NCT05920967
Title: Effect of Continuous Paravertebral Nerve Block Combined With Dexamethasone Palpitate vs Combined With Dexamethasone Sodium Phosphate on Chronic Postoperative Pain in Patients Undergoing Minimally Invasive Cardiac Surgery
Brief Title: PANDORA: Paravertebral AdjuNctive DexamethasOne Palmitate Reducing Chronic Pain After Caridiac Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Clinical Professor, Xijing Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20232194-C-1
Record Dates: First submitted 2023-06-15; First posted 2023-06-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — dexamethasone 21-palmitate; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DXP group (Experimental): The participants in DXP group will receive a first dose of a single paravertebral space infusion of 21 ml of analgesic containing 0.5 percentage ropivacaine 20 ml and dexamethasone palmitate 1ml.
  Interventions: Drug: Dexamethasone Palmitate
- DXM group (Active Comparator): The participants in DXM group will receive a single infusion of a paravertebral space first dose of 21 ml of analgesic containing 0.5 percentage ropivacaine 20 ml and dexamethasone sodium phosphate 1ml.
  Interventions: Drug: Dexamethasone Sodium Phosphate

INTERVENTIONS:
Drug: Dexamethasone Palmitate — a single paraverteal space infusion of 21 ml of the first dose of analgesia, consisting of 0.5 percentage ropivacaine 20 ml and dexamethasone palmitate 1ml. Then, a continuous paraverteal nerve block pump was connected for postoperative analgesia. The liquid of the pump was 250 ml 0.2 percentage ropivacaine. The background of the pump was set to 5 ml/h and PCA was set to 5 ml at an interval of 30 min.
  Arms: DXP group
Drug: Dexamethasone Sodium Phosphate — a single paraverteal space infusion of 21 ml of the first dose of analgesia, consisting of 0.5 percentage ropivacaine 20 ml and dexamethasone sodium phosphate 1ml. Then, a continuous paraverteal nerve block pump was connected for postoperative analgesia. The liquid of the pump was 250 ml 0.2 percentage ropivacaine. The background of the pump was set to 5 ml/h and PCA was set to 5 ml at an interval of 30 min.
  Arms: DXM group

SUMMARY:
The goal of this single-center, prospective, double-blind randomized controlled clinical trial is to explore preventive interventions for chronic postoperative pain (CPSP) in patients undergoing minimally invasive cardiac surgery. The main questions it aims to answer is: the incidence of CPSP is high and severe, and there is no safe and effective method for prevention and treatment. The participants in the dexamethasone palmitate (DXP) group will receive a single paravertebral space infusion of 21 ml of the first dose of analgesia, consisting of 0.5 percentage ropivacaine 20 ml and dexamethasone palmitate 1ml. The participants in dexamethasone sodium phosphate (DXM) group will receive a single infusion of a paravertebral space first dose of 21 ml of analgesic containing 0.5 percentage ropivacaine 20 ml and dexamethasone sodium phosphate 1ml. Then both groups use a continuous paravertebral nerve block pump for postoperative analgesia. The liquid of the pump is 250 ml 0.2 percentage ropivacaine. The background of the pump is set to 5 ml/h and PCA is set to 5 ml at an interval of 30 min.

DETAILED DESCRIPTION:
Minimally invasive cardiac surgery has the advantages of small injury, rapid recovery and international leadership. But the incidence of chronic pain after operation is high, which is reported to be as high as 70 percentage in thoracic intercostal surgery, seriously affecting the quality of life of patients after surgery. Uncontrolled acute pain after surgery poses the greatest risk factor for CPSP. Procedure-specific postoperative pain management (PROSPECT) guidelines recommend that the use of paravertebral nerve block as the first choice for multimodal analgesia in intercostal surgery can significantly reduce the incidence of postoperative acute pain. But there is not enough evidence to prove that it can reduce the incidence of CPSP. Choosing a reasonable combination of analgesics in nerve block to inhibit the production and transmission of multi-source nociceptive signals caused by intercostal nerve injury and inflammatory stimulation is one of the research hotspots to prevent the transformation from acute pain to chronic pain.

Dexamethasone can play an anti-inflammatory effect by reducing the sensitivity caused by neuroinflammation, which has also been confirmed by small sample studies. But a large number of literatures point out that a single use of dexamethasone cannot significantly reduce the incidence of CPSP. This may be due to the fact that the half-life of dexamethasone is only 48 hours, and single use is not enough to exert anti-inflammatory effects; long-term large-scale use can increase blood sugar concentration, leading to complications such as poor wound healing. From this, the investigators infer that finding a means or preparation to prolong the action time and efficacy of dexamethasone while reducing side effects may become an important means of preventing CPSP.

Dexamethasone palmitate is a kind of dexamethasone nanoparticles with long curative effect, good effect and few side effects. It plays a very significant therapeutic role in the late stage of inflammation and has been proved to prevent the progression of inflammation. And there have been studies on the injection of dexamethasone palmitate in epidural or perineural space, but the safety and efficacy of dexamethasone palmitate in paravertebral space need to be further studied.

The primary aim of this study is to compare whether single injection of dexamethasone palmitate and dexamethasone sodium phosphate around the paravertebral nerve combined with continuous paravertebral nerve block for postoperative analgesia can reduce the incidence of chronic pain 3 months after operation.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA class I-III
2. 18 years to 65 years
3. Undergoing intercostal incision cardiac surgery

Exclusion Criteria:

1. Urgent surgery
2. BMI≧35kg/m^2
3. Non-first cardiac surgery
4. Local anesthetic allergy
5. Skin damage or infection at the puncture site
6. Dysfunction of liver, kidney and blood coagulation
7. Previously had chronic pains

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic postoperative pain | 3 months after surgery
  Pain status score on the Brief Pain Inventory（BPI-NRS score range, 0-10; ≥1 indicates it happens）

SECONDARY OUTCOMES:
Morphine consumption | 24, 48, 72 hours after surgery
  Total consumption of rescue analgesia by oral morphine equivalent (mcg/kg)
The incidence of acute pain at resting and activity | 24, 48, 72 hours after surgery
  Numerical Rating Scale to evaluate the incidence of pain (NRS score range, 0-10; ≥1 indicates it happens once)
The incidence of chronic postoperative pain | 6 and 12 months after surgery
  Pain status score on the Brief Pain Inventory（BPI-NRS score range, 0-10; ≥1 indicates it happens）
Pain severity in the past 7 days | 3, 6, 12 months after surgery
  Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v2.0 - Pain Intensity 3a (T-score range, 36.3-81.8; 81.8 indicates worst pain intensity)
Pain severity in the past 24 hours | 3, 6, 12 months after surgery
  Brief Pain Inventory (BPI pain intensity score rang, 0-40; 40 indicates worst pain intensity)
The interference of chronic postoperative pain on activities of daily living in the past 7 days | 3, 6, 12 months after surgery
  PROMIS Short Form v1.1 - Pain Interference 8a (PROMIS-PI-SF-8A; T-score range, 40.7-77; 77 indicates worst pain interference)
The interference of chronic postoperative pain on activities of daily living in the past 24 hours | 3, 6, 12 months after surgery
  Brief Pain Inventory (BPI pain interference score rang 0-70; 70 indicates worst pain interference)
The impact of chronic postoperative pain on neuropathic pain | 3, 6, 12 months after surgery
  PROMIS Scale v2.0 - Neuropathic Pain Quality 5a (T-score range, 37.0-74.1; 74.1 indicates highly neuropathic pain)
The impact of chronic postoperative pain on health related quality of life | 3, 6, 12 months after surgery
  12-item Short-Form Health Survey v2 (SF-12 v2.0 scores range, 0-100, 100 indicates best functioning)
The impact of chronic postoperative pain on sleep quality | 3, 6, 12 months after surgery
  Pittsburgh Sleep Quality Index (PSQI score range, 0-21, 21 indicates worst sleep quality)
The impact of chronic postoperative pain on emotional wellbeing | 3, 6, 12 months after surgery
  Hospital Anxiety and Depression Scale (HADS score range, 0-21, 21 indicates worst anxiety or depression)
The impact of chronic postoperative pain on self-efficacy | 3, 6, 12 months after surgery
  Pain Self Efficacy Questionnaire (PSEQ score range, 0-60, 60 indicates strongest self-belief)

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, MD&phD, Principal Investigator — Xijing Hospital; Taoyuan Zhang, M.D., Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, China

REFERENCES:
- [Derived] Zhang H, Zhang T, Zheng Z, Gao J, Gao B, Hou L, Zhao J, Wang L, Dong H, Lei C. Rationale and design for the thoracic Paravertebral Adjunctive Dexamethasone Palmitate Reducing chronic pain After cardiac surgery (PANDORA) trial: a parallel-group, double-blinded, randomised controlled, single-centre study. BMJ Open. 2025 Jan 15;15(1):e086392. doi: 10.1136/bmjopen-2024-086392. PMID 39819928